CLINICAL TRIAL: NCT06181409
Title: Diagnosing and Monitoring Portal Hypertension Non-invasively Using Spleen Stiffness Measurement in Patients With Advanced Chronic Liver Disease: a Prospective Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Amine Benmassaoud, Division of Gastroenterology and Hepatology Assistant Professor of Medicine, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: MP-2022-8165
Record Dates: First submitted 2023-12-01; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Advanced Chronic Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to assess non-invasive tools' efficacy in predicting portal hypertension-related complications in individuals with advanced chronic liver disease. The main question it aims to answer are:

- what are the cut-off values for non-invasive tests (NITs) (including LSM, SSM) that predict the presence and occurrence of hepatic decompensation in individuals with advanced chronic liver disease?

Participants will undergo regular study visits involving non-invasive tests (LSM, SSM) and assessments to monitor hepatic decompensation over the study period.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18years old
* Advanced chronic liver disease (defined as LSM ≥ 10kPa)
* Ability to provide informed consent

Exclusion Criteria:

* Transjugular intrahepatic portosystemic shunt
* previous liver transplantation
* Abnormality of the porto-mesenteric system (portal vein thrombosis, splenic vein thrombosis, splenectomy, portal cavernomatous transformation, porto-caval shunts)
* Hematological malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with advanced chronic liver disease (defined as LSM ≥ 10kPa)
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients diagnosed with portal hypertension using elastography techniques | At baseline
  We will assess the diagnostic accuracy of liver and spleen stiffness for portal hypertension

SECONDARY OUTCOMES:
Identifying patients at high-risk of liver related events using elastography techniques | 5 years
  We will use liver and spleen stiffness to identify patients at risk of developing liver -related events

IPD SHARING:
Plan to Share IPD: No